CLINICAL TRIAL: NCT02652169
Title: Platelet Rich Fibrin in Combination With Topical Antibiotics or Antiseptics in the Treatment of Chronic Wounds - a Prospective, Randomized, Active Controlled, Double Blind Pilot Trial With an Observer-blinded Control Group
Brief Title: PRF With Topical Antibiotics or Antiseptics in Chronical Wounds Version 1.4
Acronym: PRF-TAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, Univ.-Prof. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRF-TAT
Record Dates: First submitted 2015-07-17; First posted 2016-01-11 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Chronic Skin Ulcer
MeSH Terms: interventions — Amikacin; Teicoplanin; Prolactin-Releasing Hormone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study arm 1 - PRF plus amikacin and teicoplanin (Experimental): PRF mixed with amikacin and teicoplanin is sprayed on the patients' ulcer
  Interventions: Drug: PRF mixed with amikacin and teicoplanin
- Study arm 2 - PRF plus normal saline (Experimental): PRF mixed with normal saline is sprayed on the patients' ulcer
  Interventions: Drug: PRF plus normal saline
- Study arm 3 - PRF mixed with PHMB plus Macrogolol (Experimental): PRF mixed with polyhexanide and macrogolol is sprayed on the patients' ulcer
  Interventions: Drug: PRF mixed with PHMB plus Macrogolol
- Study arm 4 - Acticoat 7 (Active Comparator): A silver gauze (Acticoat 7®) is applied to the patients' ulcer
  Interventions: Other: Silver gauze

INTERVENTIONS:
Drug: PRF mixed with amikacin and teicoplanin — PRF, mixed with amikacin and teicoplanin is applied to the chronic ulcer
  Other Names: PRF plus amikacin/teicoplanin
  Arms: Study arm 1 - PRF plus amikacin and teicoplanin
Drug: PRF mixed with PHMB plus Macrogolol — PRF, mixed with Lavasorb is applied to the chronic ulcer
  Other Names: PRF plus Lavasorb
  Arms: Study arm 3 - PRF mixed with PHMB plus Macrogolol
Drug: PRF plus normal saline — PRF as a monosubstance plus sodium chloride 0.9% is applied to the chronic ulcer
  Other Names: PRF plus sodium chloride 0.9%
  Arms: Study arm 2 - PRF plus normal saline
Other: Silver gauze — Acticoat 7 silver wound dressing is applied to the chronic ulcer
  Other Names: Acticoat 7
  Arms: Study arm 4 - Acticoat 7

SUMMARY:
Platelet rich fibrin (PRF) is a new therapy option for chronic wounds with yet unproven therapeutic efficacy. This randomised controlled trial aims to provide evidence of the efficacy of PRF as monotherapy as well as a growth promoting carrier matrix for antimicrobial compounds. The investigators therefore designed a four armed trial with three PRF arms which are compared to each other as well as to an active comparator. The treatment arms are as follows:

Study arm 1: PRF with amikacin and teicoplanin Study arm 2: PRF with placebo (0.9% sodium chloride) Study arm 3: PRF with PHMB (polyhexanid) plus Macrogolol (Lavasorb®) Study arm 4: Acticoat 7® wound dressing as active control Patients with infected chronic wounds may be included in this trial. Infection shall be diagnosed by an experienced senior infectious diseases specialist. Patients with untreated peripheral vascular occlusive disease as defined by an ABI (ancle brachial index) of < 0,7 are excluded from the trial as are patients with an uncontrolled diabetes mellitus or patients who have not received sufficient treatment for a diabetic foot syndrome. Any underlying illness will be treated following standard of care. In case of chronic venous insufficiency four-layered compression bandages will be applied each visit if tolerated by the patient. Alternatively compression stockings (Class III) are permitted. This is mentioned as "Disease specific treatment" in the protocol.

Patients will receive treatment for 56 days. After 28 and 56 days the wound surface will be compared to the baseline. Infection parameters (c-reactive protein and leucocyte count) will be measured weekly. Evaluation of systemic antimicrobial therapy will be performed at each visit. Systemic antimicrobial therapy is started at the discretion of a senior infectious diseases specialist.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged over 18 who are able to give informed consent
* Chronic venous ulcer with localized non-systemic soft-tissue infection diagnosed by senior infectious diseases specialist based on US FDA Guidance for Industry Chronic cutaneous ulcer and burn wounds June 2006:

  * slough and necrotic tissue
  * exsudate
  * smell
  * inflammation
  * presence of granulation tissue
  * pain
* Wound size ≥ 5 cm2 and < 200 cm2

Exclusion Criteria:

* Non-treated diabetes mellitus, HbA1c > 12 mg/dl
* Non treated (orthopaedic shoe) diabetic foot syndrome
* ABI < 0,7
* Wound size 15 cm2 and > 200 cm2
* CRP > 5 mg/dl
* Leucocytes > 15.000 /μl
* Infection of another site
* Infection of the ulcer with a pathogen with inherent resistance to amikacin and teicoplanin
* Known osteomyelitis
* Known erysipelas
* Known phlegmon
* Complicated deep tissue infection not solely treatable with PRF plus antimicrobial therapy in the opinion of a senior infectious diseases specialist
* Planned systemic antimicrobial therapy
* Active viral hepatitis (A/B/C) or active HIV infection or active syphilis
* Increased sensitivity to amikacin or teicoplanin, PHMB or macrogolol
* Increased sensitivity to tramexanic acid or batroxobin
* Presence of neoplastic growth in the ulcer
* Thrombocytopenic patients (<150.000 G/L)
* Haemoglobin < 95 g/L
* Known pregnancy or lactation
* Severe renal impairment (creatinine clearance <30 ml/min)
* History or clinical signs of impairment of the cochlea or vestibularis system
* Neuromuscular diseases (i.e. Myasthenia gravis, Parkinson's disease)
* Aminoglycoside treatment less than four weeks before inclusion
* Other reasons opposing the study participation on the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2025-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
reduction in wound area | day 56

SECONDARY OUTCOMES:
Number of patients in necessity to initiate systemic antimicrobial therapy based on the opinion of a senior infectious disease consultant arises (subjective assessment based on wound inflammation, serum c-reactive protein levels and leucocyte count) | day 0, 7, 14, 21, 28, 35, 42, 49, 56
Elevation of C-reactive protein over 7 mg/dl (normal value 0.5 mg/dl) | day 0, 7, 14, 21, 28, 35, 42, 49, 56
time to sterility of the wound | day 0, 7, 14, 21, 28, 35, 42, 49, 56
Relative wound volume and wound area reduction | on day 28 and 56
Occurrence of drug resistant bacteria in the wound | day 0, 7, 14, 21, 28, 35, 42, 49, 56
Occurrence of drug resistant bacteria in a swab of the tissue surrounding the wound or a Z-swab of the torso | on day 28 and 56

CONTACTS AND LOCATIONS:
Overall Officials: Florian Thalhammer, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided